CLINICAL TRIAL: NCT07181798
Title: Evaluation of Cervical Position and Movement Sense Using Computer Vision Technology in Healthy Individuals
Brief Title: Evaluation of Cervical Position and Movement Sense Using a Novel Computer Vision-Based Software
Status: Not yet recruiting | Type: Observational
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Collaborators: Health Institutes of Türkiye (Unknown)
Responsible Party: Principal Investigator, Mustafa Güven, Lecturer and PhD Student, Principal Investigator, Kutahya Health Sciences University
Other Study IDs: NEVSEHIRHBVU-KMYO-MG-001
Record Dates: First submitted 2025-05-18; First posted 2025-09-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cervical Proprioception
Keywords: Proprioception; Computer-Assisted Image Interpretation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteer Cohort: A single cohort of 74 healthy adult volunteers will undergo an observational test-retest reliability study of four cervical proprioception assessments using computer-vision tracking. No medical interventions will be administered.
  Two distinct assessment protocols control for learning effects and follow literature-based retest intervals:
  Protocol A (n=37): Cervical Movement Sense Target Tracking at baseline and again after one week to assess longer-term reliability.
  Protocol B (n=37): Head Relocation Test in 32 participants at baseline and again after one hour. Cervical Movement Sense Patterned Tracking and Cervical Proprioceptive Function Test in all 37 participants at baseline and again after one hour to minimize short-term learning effects. Separate participant groups prevent cross-test learning, and retest intervals (1 hour vs. 1 week) align with prior studies.

SUMMARY:
This observational study evaluates cervical proprioception using a computer vision-based system developed with OpenCV and MediaPipe. Healthy adults will perform a series of head movements while their nose tip is tracked by a camera. The primary objective is to assess the accuracy of neck position and movement perception. Data will be analyzed to determine the reliability of the tracking system. The study is non-invasive, involves no interventions, and poses minimal risk to participants. Findings may support the development of accessible diagnostic tools for clinical and research applications.

DETAILED DESCRIPTION:
This study aims to assess the test-retest reliability of computer-based cervical proprioception evaluations in healthy adults using OpenCV and MediaPipe for motion tracking. Participants will be seated in a controlled environment with a computer screen at eye level. The following four evaluations will be conducted:

Cervical Joint Position Sense (Head Relocation Error): Participants attempt to reposition their head to a perceived neutral position after flexion, extension, and rotation movements. The software records the deviation in pixels between actual and perceived head positions. Six trials per movement direction will be performed, with retesting after one hour.

Cervical Movement Sense - Patterned Tracking: Participants trace on-screen shapes (e.g., F8, ZZ) with their nose tip to evaluate movement accuracy. The total deviation from the ideal path in pixels will be measured. One practice trial and recorded attempts will be conducted, with retesting after one hour.

Cervical Movement Sense - Target Tracking: Participants follow a moving on-screen target with their nose tip. Tracking accuracy and time spent inside the target will be recorded. Three trials will be performed, with retesting after one week.

Sensorimotor Control Assessment: Participants align their head with randomly appearing visual targets for one minute. Performance will be evaluated based on the number of correct alignments and response accuracy. Three trials will be conducted, with retesting after one hour.

All data will be anonymized and analyzed for reliability using Intraclass Correlation Coefficient (ICC), Standard Error of Measurement (SEM), and Minimal Detectable Change (MDC). This non-invasive, computer-based methodology aims to provide a reliable and low-cost approach to assessing cervical joint position sense, movement perception, and sensorimotor control, contributing to future clinical and research applications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals over 18 years of age
* No neck pain

Exclusion Criteria:

* Neck or spinal symptoms
* History of cervical/spinal trauma or surgery
* Chronic conditions affecting mobility
* Visual or vestibular impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of healthy adult volunteers aged 18 years and older, without any history of neck pain, spinal disorders, or other conditions affecting cervical mobility. Participants will be recruited from the general population.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cervical Joint Position Sense (Head Relocation Error) | The test will be repeated at 1-hour intervals.
  With the help of algorithms, the initial position of the participant's nose tip on the screen will be recorded. Following flexion, extension, or rotation movements, the final position will be obtained, and the difference between the initial and final positions will be calculated in pixels and reported as the error score. While the primary output will be in pixels, this difference can also be expressed in degrees with the necessary conversions. Rotational movements performed during the measurement will be simultaneously recorded using the CROM device, and the values from the screen will be compared with those from the CROM to assess criterion validity, which provides the error magnitude directly in degrees. Measurements performed on the same group at two different time points will be analyzed using the Intraclass Correlation Coefficient (ICC), the Standard Error of Measurement (SEM), and Bland-Altman methods.
Cervical Movement Sense - Patterned Tracking | The test will be repeated at 1-hour intervals.
  During the test, an F8 or ZZ shaped pattern will be displayed on the screen, and the participant will trace the pattern starting from the center using their nose tip. The algorithm will track the nose tip's position in each camera frame throughout the test: if the nose tip remains within the shape, the error score will be 0; if it moves outside, the distance to the nearest point of the shape will be calculated in pixels and recorded as the instantaneous error score. At the end of the test, all instantaneous error scores will be summed to obtain the total error score. The start and finish times of the test will also be recorded to determine the total test duration. Total error scores from measurements performed on the same group at different time points will be analyzed using the Intraclass Correlation Coefficient (ICC), the Standard Error of Measurement (SEM), and Bland-Altman methods.
Cervical Movement Sense - Target Tracking: | The test will be repeated at 1-week intervals.
  During the test, a rectangle will appear on the screen and move at a constant speed along the ZZ or F8 paths. The participant will attempt to keep their nose tip inside this moving rectangle. Since the speed is fixed, the test duration is the same for all participants.
  Scoring Methods
  Time-Based Score: The total time the nose tip remains inside the rectangle is divided by the total test duration. The resulting ratio ranges from 0 to 1:
  1 → Best score (nose tip always inside)
  0 → Worst score (nose tip never inside)
  Distance-Based Score: For each frame, the algorithm calculates the distance from the nose tip to the rectangle:
  Inside = 0
  Outside = distance in pixels to the nearest edge
  At the end, all distances are summed to obtain the total deviation score. Both scores from measurements performed on the same group at different time points will be analyzed using the Intraclass Correlation Coefficient (ICC), the Standard Error of Measurement (SEM), and Bland-Altman methods.
Sensorimotor Control Assessment | The test will be repeated at 1-hour intervals.
  The test duration is 60 seconds. During this time, individual points will appear on the screen at random locations.
  The participant's task is to move their nose tip over these points. When the nose tip correctly reaches a point:
  The point will disappear,
  A new point will appear at a different location on the screen.
  At the end of the test, the number of points the participant successfully matched with their nose tip within the 60 seconds will be counted, and this value will be recorded as the test score.
  The test score obtained from measurements performed on the same group at different time points will be analyzed using the Intraclass Correlation Coefficient (ICC), the Standard Error of Measurement (SEM), and Bland-Altman methods.

CONTACTS AND LOCATIONS:
Overall Officials: ismail Saraçoğlu, Associate Professor, Principal Investigator — Kütahya University of Health Sciences
Locations (1):
- Nevşehir Hacı Bektaş Veli University, Nevşehir, Kozakli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zou GY. Sample size formulas for estimating intraclass correlation coefficients with precision and assurance. Stat Med. 2012 Dec 20;31(29):3972-81. doi: 10.1002/sim.5466. Epub 2012 Jul 4. PMID 22764084
- [Background] Mondal D, Vanbelle S, Cassese A, Candel MJ. Review of sample size determination methods for the intraclass correlation coefficient in the one-way analysis of variance model. Stat Methods Med Res. 2024 Mar;33(3):532-553. doi: 10.1177/09622802231224657. Epub 2024 Feb 6. PMID 38320802
- [Background] Basteris A, Pedler A, Sterling M. Evaluating the neck joint position sense error with a standard computer and a webcam. Man Ther. 2016 Dec;26:231-234. doi: 10.1016/j.math.2016.04.008. Epub 2016 Apr 23. PMID 27161883
- [Background] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Background] Sarig-Bahat H, Weiss PL, Laufer Y. Cervical motion assessment using virtual reality. Spine (Phila Pa 1976). 2009 May 1;34(10):1018-24. doi: 10.1097/BRS.0b013e31819b3254. PMID 19404177
- [Background] Pinsault N, Fleury A, Virone G, Bouvier B, Vaillant J, Vuillerme N. Test-retest reliability of cervicocephalic relocation test to neutral head position. Physiother Theory Pract. 2008 Sep-Oct;24(5):380-91. doi: 10.1080/09593980701884824. PMID 18821444
- [Background] Strimpakos N, Sakellari V, Gioftsos G, Kapreli E, Oldham J. Cervical joint position sense: an intra- and inter-examiner reliability study. Gait Posture. 2006 Jan;23(1):22-31. doi: 10.1016/j.gaitpost.2004.11.019. PMID 16311191
- [Background] Werner IM, Ernst MJ, Treleaven J, Crawford RJ. Intra and interrater reliability and clinical feasibility of a simple measure of cervical movement sense in patients with neck pain. BMC Musculoskelet Disord. 2018 Oct 5;19(1):358. doi: 10.1186/s12891-018-2287-0. PMID 30290759
- [Background] Kristjansson E, Oddsdottir GL. "The Fly": a new clinical assessment and treatment method for deficits of movement control in the cervical spine: reliability and validity. Spine (Phila Pa 1976). 2010 Nov 1;35(23):E1298-305. doi: 10.1097/BRS.0b013e3181e7fc0a. PMID 20975484
- [Background] Kristjansson E, Hardardottir L, Asmundardottir M, Gudmundsson K. A new clinical test for cervicocephalic kinesthetic sensibility: "the fly". Arch Phys Med Rehabil. 2004 Mar;85(3):490-5. doi: 10.1016/s0003-9993(03)00619-1. PMID 15031839
- [Background] Hage R, Ancenay E. Identification of a relationship between cervical spine function and rotational movement control. Ann Phys Rehabil Med. 2009 Nov;52(9):653-67. doi: 10.1016/j.rehab.2009.04.003. Epub 2009 Sep 10. English, French. PMID 19783494
- [Background] Goncalves C, Silva AG. Reliability, measurement error and construct validity of four proprioceptive tests in patients with chronic idiopathic neck pain. Musculoskelet Sci Pract. 2019 Oct;43:103-109. doi: 10.1016/j.msksp.2019.07.010. Epub 2019 Jul 28. PMID 31376618
- [Background] English DJ, Zacharias A, Green RA, Weerakkody N. Reliability of Cervicocephalic Proprioception Assessment: A Systematic Review. J Manipulative Physiol Ther. 2022 Jun;45(5):346-357. doi: 10.1016/j.jmpt.2022.08.005. Epub 2022 Oct 19. PMID 36270904
- [Background] Sarig Bahat H, Sprecher E, Sela I, Treleaven J. Neck motion kinematics: an inter-tester reliability study using an interactive neck VR assessment in asymptomatic individuals. Eur Spine J. 2016 Jul;25(7):2139-48. doi: 10.1007/s00586-016-4388-5. Epub 2016 Jan 30. PMID 26831536